CLINICAL TRIAL: NCT02476682
Title: Evaluation of Stool and Blood Based Tests for Colorectal Advanced Mucosal Neoplasia
Brief Title: Non-invasive Risk Stratification of CR AMN/SSP
Acronym: FIT
Status: Terminated | Type: Observational
Why Stopped: facility required for analysis of samples is no longer able to facilitate analysis
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2014/9/4.4(4079)
Record Dates: First submitted 2015-06-10; First posted 2015-06-19 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Adenomatous Polyps
Keywords: Sessile serrated polyps; Advanced mucosal neoplasia
MeSH Terms: conditions — Adenomatous Polyps | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2mg of stool per patient 18mL of blood per patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Normal subjects: blood or stool samples will be collected from people referred for screening colonoscopy
  Interventions: Other: blood or stool samples will be collected
- Colorectal cancer: blood or stool samples will be collected from people with colorectal cancer detected at colonoscopy or resection
  Interventions: Other: blood or stool samples will be collected
- Polyps <10mm and no high risk features: blood or stool samples will be collected from people with no polyps or low risk polyps (<10mm, no villous component or dysplasia) detected at colonoscopy
  Interventions: Other: blood or stool samples will be collected
- Advanced Mucosal Neoplasia: blood or stool samples will be collected from people with AMN detected at resection
- Sessile Serrated Adenoma: blood or stool samples will be collected from people with SSP detected at resection
- non-colorectal neoplastic disease: Participants with disease that is not colorectal neoplasia. Analysis of this cohort is not a primary endpoint but the investigators will report assay positivity in this group on an opportunistic basis. This cohort will include patients diagnosed with, for example, inflammatory bowel disease or extracolonic cancer.
  Interventions: Other: blood or stool samples will be collected

INTERVENTIONS:
Other: blood or stool samples will be collected — blood or stool samples will be collected
  Groups: Colorectal cancer; Normal subjects; Polyps <10mm and no high risk features; non-colorectal neoplastic disease

SUMMARY:
The purpose of this study is to determine the clinical utility of stool and blood methylation tests for detection of advanced mucosal neoplasia (AMN) and sessile serrated polyps (SSP).

DETAILED DESCRIPTION:
By not only diagnosing colorectal cancer (CRC) at an early stage, but also removing precursor lesions (adenomas), colonoscopy with polypectomy reduces the risk of developing and dying from CRC. Approximately 90% of polyps are less than 10 mm and are easily removed by competent endoscopists. Laterally spreading lesions (LST) and sessile lesions of the colon, also known as advanced mucosal neoplasia (AMN) are underrecognised types of lesions that are more likely to progress to cancer. They include sessile serrated polyps (SSP), an emerging entity of flat polyps with malignant potential. Detection of hemoglobin (a component of blood) in stool is an established validated screening tool for CRC. Its specific role in the prediction of AMN, and particularly SSPs is yet to be defined. Blood tests measuring the level of tumour derived methylated deoxyribonucleic acid (DNA) in blood circulating have been demonstrated to have clinical utility for detection of CRC and AMN. A blood based CRC screening test has the potential to increase compliance. This study aims to determine the clinical utility of stool and blood methylation tests for detection of AMN and SSPs. Stool and blood will be obtained from consenting patients referred for endoscopic removal of known ANM and SSP (study arm) as well as from consenting patients scheduled for colonoscopy screening (control arm). The level of stool hemoglobin and methylated tumour derived DNA in circulation will be measured in the two study groups. Cutoff values will be generated to assess best predictive capability of high risk lesions based on these tests.

ELIGIBILITY:
Inclusion Criteria:

* Individuals capable and willing of proving satisfactory informed consent
* Individuals with colonic lesions larger than 20mm
* Individuals diagnosed with laterally spreading or sessile polyp morphology
* Individuals schedules for screening colonoscopy and with no prior history of CRC
* Ability and willingness to collect stool sample at home
* Ability and willingness to undergo venepuncture procedure

Exclusion Criteria:

* Individuals not able or unwilling to provide informed consent
* Individuals less than 18 year of age
* Individuals who undergo an incomplete colonoscopy or resection, which raises doubt as to the status of the colon (post-hoc exclusion)
* Individuals with a prior history of CRC
* Individuals with a history of Irritable Bowel Disease (IBD), hereditary nonpolyposis colorectal cancer (HNPCC) or Familial adenomatous polyposis (FAP)
* Individuals with bleeding diathesis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of subjects diagnosed with AMN/SSP and subjects scheduled for screening colonoscopy.
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Demographics | 1 day
  Data to adequately describe demographic situations of each participant.
Level of methylated DNA in circulation | 5 years
  The process will use an automated extraction procedure incorporating state-of-the-art magnetic silica-coated beads on a QIASymphony (Qiagen). The extracted DNA is bisulphite-converted and further purified (automated on a QIACube HT liquid handler) prior to analyzing 12uL of bis-DNA in a multi-plexed (BCAT1, IKZF1, ACTB (control assay)) real-time PCR for measuring the methylation levels of target amplicons.
Level of haemoglobin in stool | 5 years
  Suspended stool collected in the HM-JACKarc sampling device will be processed for Hb measurements using commercially available reagents and the bench-top analyser instrument, HM-JACKarc, according to manufacturer recommendation (Kyowa Medex Co Ltd, Japan). Measured haemoglobin concentrations will be reported as ug Hb/g stool. A 20 ug Hb/g stool a cut-off concentration will be used for qualitative reporting.
Demographics | 1 day
  Data to adequately decribe the clinical situations of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS FRACP, Principal Investigator — Westmead Hospital
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia